CLINICAL TRIAL: NCT04675905
Title: Patient-Centred Outcomes and Resource Utilisation After Noncardiac Surgery-D(Eutschland) (PACORUS-D)
Acronym: PACORUS-D
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PD Dr. med. MSc Giovanna Lurati Buse (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other); University Hospital, Bonn (Other); University Hospital, Aachen (Other); University Hospital of Cologne (Other); University Hospital, Essen (Other); University Hospital Heidelberg (Other); Ruhr University of Bochum (Other); German Society of Anesthesiology and Intensive Care (DGAI) (Unknown)
Responsible Party: Sponsor-Investigator, PD Dr. med. MSc Giovanna Lurati Buse, Principal Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: PACORUS-D
Record Dates: First submitted 2020-12-10; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Noncardiac Surgery
Keywords: Outcome Assessment, Health Care [Mesh];; Surgical Procedures, Operative, Economics; noncardiac surgery; disability; patient-centred outcome
MeSH Terms: interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PACORUS-D Main cohort: Eligibility, Endpoints as described above
  Interventions: Other: no intervention (cohort study)
- PACORUS-D Delirium-Subcohort: Eligibility: patients aged >= 65 years undergoing noncardiac nonneurosurgical procedures (definition see above); Endpoints as described above; additional explanatory variable: postoperative Delirium detected by CAM on postoperative day 1 and 2
  Interventions: Other: no intervention (cohort study)

INTERVENTIONS:
Other: no intervention (cohort study) — Explanatory variables include preoperative comorbidities, baseline disability, surgical risk, postoperative complications, sex, rural/urban area of residency, Oslo Social Support Scale; Clinical Frailty Scale in patients aged >= 65 years

SUMMARY:
The PACORUS-D project aims at 1) quantifying the 30-days and 1-year disability burden (assessed using the 12-item WHODAS 2 [WHO Disability Assessment Schedule] questionnaire) after inhospital noncardiac nonneurosurgical procedures ; 2) quantifying the resource utilization up the 1 year after inhospital noncardiac nonneurosurgical procedures; 3) validating days alive and out of hospital (construct and criterion validity) in Germany. PACORUS-D consists of 2 independent cohort: a clinical multicentre cohort to assess "disability" and "days alive and out of hospital" and an administrative cohort to assess "days alive and out of hospital" and "resource utilization" from statutory health insurance data. PACORUS-D is intended as preparatory project in Germany before international expansion. THIS REGISTRATION REFERS TO THE CLINICAL COHORT ONLY.

DETAILED DESCRIPTION:
Objectives:

1a) to quantify patient-reported disability measured using the 12-item WHO Disability Assessment Schedule (WHODAS) after noncardiac surgery

1. b) to assess the impact of preoperative comorbidities (and frailty in patients aged ≥65 years) and procedural risk, and of postoperative complications on 365-day patient-reported disability after noncardiac surgery;
2. a) to quantify days alive and out of hospital (DAOH), a recently proposed, integrative, easily collected and statistically-efficient outcome after noncardiac surgery;

2b) to validate (construct [convergent] validity) DAOH at 30 and 365 days after noncardiac surgery, i.e. to assess impact of preoperative risk factors/procedural risk and postoperative complications on DAOH; 2c) to assess in a subcohort of patients ≥ 65 years, the construct (convergent) validity of DAOH in terms of frailty (Clinical Frailty Scale);

3a) to evaluate the criterion (concurrent) validity of DAOH for patient-reported disability at 30 days and 365 days; 3b) to evaluate the criterion (predictive) validity of DAOH at 30 days for patient-reported disability at 365 days.

In addition to the main study, patients≥ 65 years may opt to participate (separate consent) to a nested cohort study to assess the impact of delirium detected by Confusion Assessment Method (CAM) on 365-day patient-reported disability after noncardiac surgery and on DAOH.

Design:

prospective multicentre cohort with nested subcohort (Delirium)

Eligibility:

Inclusion criteria:

* aged ≥50 years
* non-cardiac, non-neurosurgical surgery (thoracic, vascular, abdominal, urinary tract, or orthopaedic/trauma)
* inhospital procedure

Patients will be excluded if:

* they are unwilling or unable to provide informed consent,
* the procedure is cancelled
* they are submitted to a procedure requiring only local anesthetics or analgosedation,
* they were submitted to ≥1 surgical procedure in the 7 days prior to enrollment
* they are unable to complete the WHODAS questionnaire (e.g. language or literacy barriers);
* they were previously enrolled in PACORUS.

Endpoints:

For objectives1a-b and 3a-b, the main endpoint will be "new onset clinically significant disability" at 365 days, defined as an increase in WHODAS score of at least 5% from baseline to a final WHODAS score of at least 35% (Shulman Anesthesiology 2020).

For objectives2a-c, the main endpoint will be days alive and out of hospital. The time horizon will be 30 days (primary) and 365 days.

Additional endpoints will include "new onset clinically significant disability" at 30 days and "clinical relevant disability" at 30 and at 365 days, defined as 12-item WHODAS exceeding 35% (Shulman Anesthesiology 2020); the continuous WHODAS score at 30 days and 365 days; disability defined at 25%.

ELIGIBILITY:
Eligibility:

Inclusion criteria:

* aged ≥50 years
* non-cardiac, non-neurosurgical surgery (thoracic, vascular, abdominal, urinary tract, or orthopaedic/trauma)
* inhospital procedure

Patients will be excluded if:

* they are unwilling or unable to provide informed consent,
* the procedure is cancelled
* they are submitted to a procedure requiring only local anesthetics or analgosedation,
* they were submitted to ≥1 surgical procedure in the 7 days prior to enrollment
* they are unable to complete the WHODAS questionnaire (e.g. language or literacy barriers);
* they were previously enrolled in PACORUS.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
New onset clinically significant disability | 365 days
  applies to objectives 1a-b and 3a-b; Definition:increase in 12-item WHO Disability Assessment Schedule (WHODAS 2) score of at least 5% from baseline to a final WHODAS score of at least 35% (Shulman Anesthesiology 2020); For calculation of the 12-item WHODAS score percentage, the ordinal categories of Linkert scale for each item will be assigned numerical values (none=0 to extreme=4) for a total maximal score of 48 and transformed into the percentage of maximal disability score (Ustun, Bull World Health Organ, 2010); higher percentage indicates higher disability.
Days alive and out of hospital | 30 days
  applies to objective 2a-c

SECONDARY OUTCOMES:
New onset clinically significant disability at 30 days | 30 days
  applies to objectives 1a-b and 3a-b; Definition see Outcome 1
Days alive and out of hospital | 365 days
  applies to objective 2a-c

OTHER OUTCOMES:
Clinical relevant disability | 30 days and 365 days
  Definition:12-item WHODAS 2 exceeding 35% (Shulman Anesthesiology 2020); for calculation of WHODAS percentage please refer to outcome 1
Continuous 12-item WHODAS 2 score | 30 days and 365 days
Disability | 30 days anf 365 days
  Definition: 12-item WHODAS 2 exceeding 25% (Ustun, Bull World Health Organ, 2010); for calculation of WHODAS percentage please refer to outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna AL Lurati Buse, MD, MSc, Principal Investigator — Anesthesiology Department, University Hospital Düsseldorf

IPD SHARING:
Plan to Share IPD: No
Pseudonymized data can not be shared due to data protection regulation. Anonymized data might be shared upon reasonable request